CLINICAL TRIAL: NCT04462419
Title: 18F-Fluciclovine PET Discrimination of Radiation Injury to the Brain
Brief Title: 18F-fluciclovine PET/MRI Imaging for the Detection of Tumor Recurrence After Radiation Injury to the Brain
Status: Terminated | Type: Observational
Why Stopped: slow enrollment
Sponsor: Mayo Clinic (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: MC1975; NCI-2020-04564 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1975 (Other: Mayo Clinic in Florida); 19-004459 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Intracranial Malignant Neoplasm; Recurrent Intracranial Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; fluciclovine F-18

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic (18F-fluciclovine, PET/MRI imaging): Patients receive fluciclovine IV and undergo brain dynamic PET/MRI imaging over 50 minutes.
  Interventions: Radiation: Dynamic Contrast-Enhanced Magnetic Resonance Imaging with Positron Emission Tomography; Other: Fluciclovine F18

INTERVENTIONS:
Radiation: Dynamic Contrast-Enhanced Magnetic Resonance Imaging with Positron Emission Tomography — Undergo PET-MRI imaging
  Other Names: DCE-MRI with PET; DCE-MRI/PET
Other: Fluciclovine F18 — Given IV
  Other Names: (18F)Fluciclovine; (18F)GE-148; 18F-Fluciclovine; [18F]FACBC; Anti-(18f)FABC; Anti-1-Amino-3-[18F]Fluorocyclobutane-1-Carboxylic Acid; Anti-[18F] FACBC; Axumin; Fluciclovine (18F); FLUCICLOVINE F-18; GE-148 (18F); GE-148 F-18

SUMMARY:
This phase I trial studies the ability and amount of fluciclovine positron emission tomography (PET) imaging needed to recognize tumors that have come back (recurrence) after brain injury from radiation therapy (radionecrosis) in patients with intracranial disease that has spread to other places in the body (metastatic). F-18 fluciclovine is a radiotracer that works by accumulating in tumor cells, making it easier to detect tumors. The results of this study may also help investigators understand all the ways that F-18 fluciclovine may affect patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the static fluciclovine F18 (fluciclovine) PET imaging tumor-to-background ratios (TBRmax; TBRmean) which distinguish true tumor recurrence from radionecrosis in patients with intracranial metastatic disease previously treated with radiation therapy, and magnetic resonance imaging (MRI) findings suggesting recurrent disease, using histopathology as proof of disease.

SECONDARY OBJECTIVES:

I. To determine static fluciclovine PET standardized uptake value (SUV)peak, SUVmean values and metabolic tumor volumes (MTV) which distinguish true tumor recurrence from radionecrosis in patients with MRI findings suggesting recurrent disease, using serial MRI as a surrogate marker of disease.

II. To determine early dynamic fluciclovine PET time activity curve values which distinguish true tumor recurrence from radionecrosis in patients with MRI findings suggesting recurrent disease, using histopathology or serial MRI as a marker of disease.

III. To correlate the determined static fluciclovine PET SUVpeak, SUVmean, TBRmax, TBRmean, and MTV values with progression free survival.

IV. In patients with true tumor progression, SUV values will be correlated with Ki67 staining on final pathology.

OUTLINE:

Patients receive fluciclovine intravenously (IV) and undergo brain dynamic PET/MRI imaging over 50 minutes.

After completion of study, patients are followed up every 3 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of intracranial metastatic disease which underwent radiation and who presents with MRI findings suspicious for recurrent disease and/or radionecrosis (namely the 'index lesion')

Exclusion Criteria:

* Contraindication to contrast enhanced MRI
* Females of child-bearing potential who are pregnant or lactating or who are not using adequate contraception (surgical, hormonal or double barrier, i.e. condom and diaphragm)
* Inability to lie still for 50 minutes during fluciclovine PET-MRI imaging
* Inability or refusal to consent
* Allergy or anaphylaxis to any of the reagents used in this study
* Inability or unwillingness to return for required visits and follow-up exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial metastatic disease (brain tumor) that has been treated with radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Tumor-to-background ratios (TBR)max and TBRmean thresholds | Up to 4 weeks post study registration
  Will be estimated to delineate tumor progression from radionecrosis for use in future studies. The optimal TBRmax and TBRmean thresholds will be chosen as the threshold with the best cutpoint/threshold during a Receiver Operating Characteristics analysis corresponding to the maximum area under the curve (AUC) value when both the sensitivity and specificity are greater than 85%.

SECONDARY OUTCOMES:
Static values for fluciclovine PET standardized uptake value (SUV)peak that distinguish true tumor recurrence from radionecrosis in patients with MRI findings suggesting recurrent disease | Up to 4 weeks post study registration
  Determined using serial MRI as a surrogate marker of disease.The optimal SUVpeak, SUVmean and metabolic tumor volumes (MTV) values will be chosen as the threshold with the best cutpoint/threshold during a Receiver Operating Characteristics analysis corresponding to the maximum AUC value when both the sensitivity and specificity are greater than 85%.
Static values for fluciclovine SUVmean that distinguish true tumor recurrence from radionecrosis in patients with MRI findings suggesting recurrent disease | Up to 4 weeks post study registration
  Determined using serial MRI as a surrogate marker of disease. The optimal SUVmean values will be chosen as the threshold with the best cutpoint/threshold during a Receiver Operating Characteristics analysis corresponding to the maximum AUC value when both the sensitivity and specificity are greater than 85%.
Static values for metabolic tumor volumes (MTV) that distinguish true tumor recurrence from radionecrosis in patients with MRI findings suggesting recurrent disease | Up to 4 weeks post study registration
  Determined using serial MRI as a surrogate marker of disease. The optimal MTV values will be chosen as the threshold with the best cutpoint/threshold during a Receiver Operating Characteristics analysis corresponding to the maximum AUC value when both the sensitivity and specificity are greater than 85%.
Incidence of adverse events | Every 3 months up to 1 year
  Will be graded using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

OTHER OUTCOMES:
Early dynamic fluciclovine PET time-activity curve values which distinguish true tumor recurrence from radionecrosis | Up to 4 weeks post study registration
  Will be chosen as the threshold with the best cutpoint/threshold during a Receiver Operating Characteristics analysis corresponding to the maximum area under the curve (AUC) value when both the sensitivity and specificity are greater than 85%.
Correlation of static fluciclovine PET SUVpeak, SUVmean, TBRmax, TBRmean, and MTV values with progression free survival | Up to 1 year after completion of PET/MR imaging
  Differences in progression free survival time between patient groups based on the determined thresholds will be analyzed via Kaplan-Meier methods.
Correlation of SUV values with Ki67 staining | Up to 4 weeks post study registration
  In patients with true tumor progression, SUV values will be correlated with Ki67 staining on final pathology. Spearman correlation analysis will be performed to determine if a relationship exists between SUV values and Ki67 staining values in patients with tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M. Trifiletti, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Kotecha R, Aboian M, Nabavizadeh SA, Parent EE, Trifiletti DM, Chao ST. Letter regarding "Contribution of PET imaging to radiotherapy planning and monitoring in glioma patients-a report of the PET/RANO group": 18F-fluciclovine and target volume delineation. Neuro Oncol. 2021 Aug 2;23(8):1408-1409. doi: 10.1093/neuonc/noab097. No abstract available. PMID 34081125
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials